CLINICAL TRIAL: NCT01534936
Title: Atypical Antipsychotics in the Treatment of Affective Symptoms of Schizophrenia in Hungary.
Acronym: AFFECT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NHU-ATC-2011/1
Record Dates: First submitted 2012-02-13; First posted 2012-02-17 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Schizophrenia; Affective Symptoms
Keywords: schizophrenia; atypical antipsychotics; depressive symptoms
MeSH Terms: conditions — Schizophrenia; Affective Symptoms; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Schizophrenic outpatients with affective symptoms.

SUMMARY:
This is a noninterventional observational study lead amongst psychiatrists, to assess the the overall status of schizophrenic outpatients with affective symptoms treated with atypical antipsychotics.

DETAILED DESCRIPTION:
Atypical antipsychotics in the treatment of affective symptoms of schizophrenia in Hungary

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenic outpatients diagnosis based on DSM -IV above 18 years of age with affective symptoms.
* Atypical antipsychotic treatment at least for a month before study inclusion.

Exclusion Criteria:

* Pregnancy.
* Hepatic disease.
* Diabetes mellitus.
* Severe cerebro- or cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Schizophrenic outpatients above 18 years of age with affective symptoms.
Sampling Method: Probability Sample
Enrollment: 2153 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline on clinical global impression scale up to 6 months of schizophrenic outpatients with affective symptoms. | 3 and 6 months
  The Clinical Global Impression Scale (CGI) is a brief clinician-rated instrument. The CGI severity of illness measure (CGI-S) is rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The CGI global improvement measure (CGI-I) is rated from 1 (very much improved) to 7 (very much worse). "0" stands for "not assessed". Means and standard deviations (SD) for CGI-S(baseline), CGI-S (1.visit) CGI-S (2.visit) and for CGI-I will be calculated.

SECONDARY OUTCOMES:
Description of the relation between and the change of affective symptoms and overall clinical status. | 3 and 6 months
Assessment of the efficacy of different atypical antipsychotics in the treatment of schizophrenia with affective symptoms measured by the difference in CGI-S (CGI severity of illness measure) and CGI-I (CGI global improvement measure). | From baseline up to 6 months
  The Clinical Global Impression Scale (CGI) is a brief clinician-rated instrument. The CGI severity of illness measure (CGI-S) is rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The CGI global improvement measure (CGI-I) is rated from 1 (very much improved) to 7 (very much worse). "0" stands for "not assessed".
Assessment of the efficacy of different atypical antipsychotics in the treatment of schizophrenia with affective symptoms measured by the difference in Raskin Scale. | From baseline up to 6 months
  Raskin scale is rated from 1 not at all to 5 very much , in three aspects: verbal report, behaviour, secondary symptoms of depression. Above 9 (the sum points) is considered moderate depression.

CONTACTS AND LOCATIONS:
Overall Officials: Attila Nemeth, MD PHD, Principal Investigator — National Center of Psychiatry; Lilla Szabo, MD, Study Chair — AstraZeneca; Alexandra Heringh, MD, Study Director — AstraZeneca
Locations (53):
- Hungary (53):
  - Research Site, Agárd
  - Research Site, Baja
  - Research Site, Barcs
  - Research Site, Berettyóújfalu
  - Research Site, Bicske
  - Research Site, Bonyhád
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Debrecen
  - Research Site, Dombóvár
  - Research Site, Dunaújváros
  - Research Site, Esztergom
  - Research Site, Érd
  - Research Site, Gyöngyös
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Hatvan
  - Research Site, Heves
  - Research Site, Hódmezővásárhely
  - Research Site, Izsófalva
  - Research Site, Jánoshalma
  - Research Site, Jászberény
  - Research Site, Kalocsa
  - Research Site, Karcag
  - Research Site, Kecskemét
  - Research Site, Kiskunhalas
  - Research Site, Kiskunmajsa
  - Research Site, Kistarcsa
  - Research Site, Kistokaj
  - Research Site, Makó
  - Research Site, Miskolc
  - Research Site, Mosonmagyaróvár
  - Research Site, Nagykanizsa
  - Research Site, Nagykálló
  - Research Site, Oroszlány
  - Research Site, Pápa
  - Research Site, Pécs
  - Research Site, Pomáz
  - Research Site, Salgótarján
  - Research Site, Sátoraljaújhely
  - Research Site, Sopron
  - Research Site, Szeged
  - Research Site, Szeghalom
  - Research Site, Szekszárd
  - Research Site, Szentendre
  - Research Site, Szentes
  - Research Site, Székesfehérvár
  - Research Site, Szigetszentmiklós
  - Research Site, Szolnok
  - Research Site, Szombathely
  - Research Site, Tószeg
  - Research Site, Vác
  - Research Site, Veszprém